CLINICAL TRIAL: NCT06681948
Title: A Randomized, Double-Blind, Placebo Parallel-Controlled, Multicenter Clinical Study for Evaluating the Efficacy, Safety and Tolerability of JT821 in the Treatment of Mild and Moderate Alzheimer's Disease
Brief Title: The Ketogenic Diet in the Treatment of Alzheimer's Disease
Acronym: JT821
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: West China Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Tianjin Huanhu Hospital (Other); Shandong Provincial Hospital (Other Government); Peking University Third Hospital (Other); Shanghai Mental Health Center (Other); Beijing Tiantan Hospital (Other); Xiangya Hospital of Central South University (Other); First Affiliated Hospital of Chongqing Medical University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Sichuan Provincial People's Hospital (Other); Brain Hospital Affiliated to Guangzhou Medical University (Unknown); Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Jianping Jia, Head of Department, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XWYY-GLST-01
Record Dates: First submitted 2024-10-20; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Alzheimer Disease
Keywords: Ketogenic Diet; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Diet, Ketogenic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketogenic diet (Experimental): The subjects initially enter the screening phase (≤ 2 weeks); following randomization, they undergo the titration period (≤ 2 weeks), gradually titrating to the maximum dose stipulated in the protocol or the maximum tolerable dose for the subject; during the treatment period (26 weeks), but if intolerance emerges during the treatment, the subject can revert to the previous tolerated dose for continued treatment.
  The dosage was titrated incrementally until reaching the maximum daily dose of 30g * 3 meals/day as stipulated in the protocol or the maximum tolerable daily dose for the subject. After entering the treatment period (from week 3 to week 28), this dose was maintained for 26 weeks.
  Interventions: Dietary Supplement: Ketogenic diet
- Control (Placebo Comparator): The subjects initially enter the screening phase (≤ 2 weeks); following randomization, they undergo the titration period (≤ 2 weeks), gradually titrating to the maximum dose stipulated in the protocol or the maximum tolerable dose for the subject; during the treatment period (26 weeks), but if intolerance emerges during the treatment, the subject can revert to the previous tolerated dose for continued treatment.
  The dosage was titrated incrementally until reaching the maximum daily dose of 30g * 3 meals/day as stipulated in the protocol or the maximum tolerable daily dose for the subject. After entering the treatment period (from week 3 to week 28), this dose was maintained for 26 weeks.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Ketogenic diet — Ketogenic diet
  Arms: Ketogenic diet
Dietary Supplement: placebo — placebo
  Arms: Control

SUMMARY:
This research is a randomized, double-blind, placebo-parallel controlled, and multi-center clinical study in China, aiming to evaluate the tolerability, efficacy, and safety of JT821 (Ketogenic Diet) in the treatment of mild to moderate Alzheimer's disease.

The ketogenic diet (KD) is a low-carbohydrate, adequate protein and high-fat diet. KD was shown to be effective in treating different neurodegenerative diseases.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multi-center clinical study planned to include 300 subjects diagnosed with mild to moderate Alzheimer's disease. The primary aim of the study is to evaluate the tolerability, efficacy, and safety of JT821 in the treatment of mild to moderate Alzheimer's disease.

Eligible patients will be randomly assigned in a 1:1 ratio to either the JT821 group or the placebo group. All subjects will undergo a 2-week product titration period based on a stable and regular anti-dementia drug treatment before entering a 26 week treatment period.

Efficacy assessments will be conducted at week 13 and week 26 during the treatment period, utilizing the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-cog) and the Mini-Mental State Examination (MMSE) to assesses the overall cognitive function of the subjects. Additionally, the Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) will evaluate daily living abilities; and the Quality of Life in Alzheimer's Disease (QOL-AD) will assess the quality of life of Alzheimer's disease patients.

Safety evaluation will include the vital signs, laboratory tests (twelve-lead electrocardiogram, fasting blood glucose, blood ketone levels (β-hydroxybutyrate), urinalysis, complete blood count, fasting lipid profile, liver and kidney function), as well as the recording of any adverse events.

Subjects may withdraw from the study at any time. If subjects experience a serious adverse event, become pregnant, are lost to follow-up, show poor adherence, or if the subject or their legal guardian actively requests to withdraw or retracts informed consent, they may be withdrawn based on the investigator's determination. The sponsor reserves the right to terminate the study at any time for special reasons (such as major safety concerns, force majeure, etc.).

A safety follow-up will be conducted two weeks after the termination of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between the ages of 50 - 85;
2. Subject must have completed the sixth grade of primary school (or its equivalent) and capable of completing the cognitive ability assessments and other tests as stipulated in the protocol;
3. Meeting the diagnostic criteria for probable AD dementia of the National Institute on Aging and the Alzheimer's Association (NIA-AA) (2011);
4. Having experienced memory decline for at least 12 months and a slow progressive trend;
5. Subject with mild to moderate disease severity, specifically those who meet the following criteria at the screening visit and baseline: 11 points ≤ Mini-Mental State Examination (MMSE) total score < 26 points (for subjects with primary school education, 11 points ≤ MMSE total score ≤ 22 points); 1 point ≤ Clinical Dementia Rating Scale (CDR) total score ≤ 2 points;
6. Total score on the Hachinski Ischemic Scale (HIS) ≤ 4 points;
7. Total score on the Hamilton Depression Scale (HAMD, 17-item version) ≤ 17 points;
8. At the screening visit or within the past 6 months, subject must undergo a brain magnetic resonance imaging (MRI) plain scan and oblique coronal hippocampal scan:

   ①Showing high likelihood of AD (Visual Rating Scale of Medial Temporal Lobe Atrophy [MTA Scale] grade: Grade 1 or higher is considered abnormal);

   ②No infarct lesions in key areas such as the thalamus, hippocampus, entorhinal cortex, parahippocampal cortex, angular gyrus, cortex, and other subcortical gray matter nuclei;

   ③The grade on the Brain White Matter Lesion Rating Scale (Fazekas Scale) ≤ 2. If the patient can provide the results of the brain MRI oblique coronal hippocampal scan that meet the protocol requirements within 6 months prior to the screening visit, it can be used as the basis for enrollment and does not need to be repeated. If the researcher is unable to determine whether the subject's condition has changed, additional brain MRI plain scan and oblique coronal hippocampal scan can be conducted prior to enrollment.
9. Female patients must be postmenopausal women (postmenopause ≥ 24 weeks), have undergone surgical sterilization, or fertile women who agree to take effective contraceptive measures during the study. Fertile women or patients with a postmenopausal period shorter than 24 weeks must undergo a urine pregnancy test during the screening period, and the result must be negative;
10. Subjects are required to be receiving stable and regular anti-dementia drug treatment for more than 1 month at the first screening;
11. The subject should have a stable and reliable caregiver who can provide care for at least 4 days per week, with at least 4 hours per day. The caregiver will assist the subject throughout the study and must accompany the subject to each study visit, ensuring sufficient interaction and communication with the subject to facilitate the researcher in completing the relevant scale evaluations.
12. Prior to the screening visit examination, the subject must sign a written informed consent form. If the subject cannot sign due to limited cognitive ability or other reasons, the signature may be left blank, and the rationale must be stated. The legal guardian should provide the reason, sign the name, date, and time in the reason description area, and also sign the name, date, and time in the legal guardian column.

Exclusion Criteria:

1. Dementia caused by other factors: vascular dementia, central nervous system infections (such as AIDS, syphilis, etc.), Creutzfeldt-Jakob disease, Huntington's disease and Parkinson's disease, Lewy body dementia, traumatic brain injury dementia, other physical and chemical factors (such as drug poisoning, alcohol poisoning, carbon monoxide poisoning, etc.), significant somatic diseases (such as hepatic encephalopathy, pulmonary encephalopathy, etc.), intracranial space-occupying lesions (such as subdural hematoma, brain tumors), endocrine system disorders (such as thyroid diseases, parathyroid diseases) and dementia caused by vitamin deficiency or any other known causes;
2. Fasting blood glucose > 7.0 mmol/L or patients previously diagnosed with diabetes;
3. Having suffered from neurological diseases other than Alzheimer's disease, including cerebrovascular diseases, neurodegenerative diseases, central nervous system infections, demyelinating diseases, movement disorders, epilepsy, spinal cord diseases, peripheral neuropathy, autonomic nervous system diseases, neuromuscular junction and muscle diseases;
4. Patients diagnosed with psychiatric conditions according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), including schizophrenia or other mental illnesses, bipolar disorder, moderate to severe depression or delirium;
5. Abnormal laboratory tests at screening visit and baseline: including liver function tests (alanine aminotransferase [ALT], aspartate aminotransferase [AST]) exceeding twice the upper limit of normal; and renal function (creatinine [Cr]) exceeding 1.5 times the upper limit of normal. Slight exceedances that are not clinically significance, as judged by the investigator, may not be excluded;
6. Fasting triglycerides ≥ 5.7 mmol/L or total cholesterol ≥ 10.34 mmol/L at the screening visit and baseline;
7. Presence any of the following infections at the screening visit:

   Positive human immunodeficiency virus antibody (HIV Ab); Positive Treponema pallidum antibody (TP Ab);
8. Other active and poorly controlled systemic severe bacterial, viral, fungal or parasitic infections (excluding fungal nail infections) that the investigator deems unsuitable for participation in this clinical study, such as sepsis, pyemia, bacteremia, and pneumonia caused by novel coronavirus infection;
9. Gastrointestinal diseases that could affect the absorption or metabolism of the investigational product as judged by the investigator, within 2 months before the screening visit;
10. Having undergone major surgeries deemed unsuitable for enrollment by the investigator within 6 months before the screening visit or those planning to undergo major surgeries during the study period (The definition of major surgeries refers to Grade 3 and Grade 4 surgeries as outlined in the "Administrative Measures for Grading of Surgeries in Medical Institutions (Trial)" implemented on December 6, 2022);
11. Patients who have suffered from malignant tumors within 3 years prior to the screening visit (excluding basal cell carcinoma of the skin that has been radically cured, squamous cell carcinoma of the skin and/or carcinoma in situ that has been radically resected);
12. Having a history of alcohol or drug abuse within 1 year prior to the screening visit;
13. Known allergy to any components of the investigational product in this study;
14. Having uncorrectable visual or auditory impairments or any other conditions that would affect the assessment of the scale;
15. Lactating women;
16. Contraindications to JT821:

Absolute contraindications:

1. Type 1 diabetes
2. Primary carnitine deficiency (Laboratory tests: Hypoglycemia with low ketone levels, elevated creatine kinase (CK), etc.)
3. Carnitine palmitoyltransferase (CPT) I and II deficiency (Laboratory tests: Hypoglycemia with low ketone levels, elevated transaminases, CK, elevated blood ammonia, tandem mass spectrometry for measurement of blood acylcarnitine profile, etc.)
4. Carnitine translocase deficiency (Laboratory tests: Hypoglycemia with low ketone levels, elevated transaminases, CK, elevated blood ammonia, tandem mass spectrometry for measurement of blood acylcarnitine profile, etc.)
5. β-Oxidation disorders (Laboratory tests: Blood glucose, electrolytes, blood lipids, coagulation, liver function, kidney function)
6. Medium-chain acyl dehydrogenase deficiency (MCAD) (Laboratory tests: Hypoglycemia with low ketone levels, elevated transaminases, CK, elevated blood ammonia, metabolic acidosis, tandem mass spectrometry for measurement of blood acylcarnitine profile, etc.)
7. Long-chain acyl dehydrogenase deficiency (LCAD) (Laboratory tests: Hypoglycemia with low ketone levels, elevated transaminases, CK, elevated creatine kinase isoenzyme (CK-MB) and lactate dehydrogenase (LDH), tandem mass spectrometry for measurement of blood acylcarnitine profile)
8. Short-chain acyl dehydrogenase deficiency (SCAD) (Laboratory tests: Tandem mass spectrometry for measurement of blood acylcarnitine profile, determination of SCAD enzyme activity)
9. Long-chain 3-hydroxyacyl-CoA deficiency (Laboratory tests: Hypoglycemia with low ketone levels, elevated transaminases, CK, elevated CK-MB and LDH, analysis of blood acylcarnitine profile, etc.)
10. Medium-chain 3-hydroxyacyl-CoA deficiency (Laboratory tests: Hypoglycemia with low ketone levels, elevated transaminases, CK, elevated CK-MB and LDH, analysis of blood acylcarnitine profile, etc.)
11. Pyruvate carboxylase deficiency (Laboratory tests: Hypoglycemia with low ketone levels, elevated transaminases, CK, elevated CK-MB and LDH, analysis of blood acylcarnitine profile, etc.)
12. Porphyria (Laboratory tests: Sunlight test of urinary porphobilinogen) Relative contraindications: (Fasting blood glucose < 2.8 mmol/L, blood ketone > 0.5 mmol/L) Patients who cannot maintain adequate nutrition (17) Any other situations that the investigator considers unsuitable for participating in this study; (18)Currently participating in other drug/device clinical trials.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale-Cognitive section(ADAS-cog) | The comparison of the baseline change values between the experimental group and the control group after 26 weeks of treatment .
  The comparison of the change values from the baseline of ADAS-cog between the experimental group and the control group after 26 weeks of treatment. ADAS-cog assesses seven aspects of cognitive function: word recall, instructions, structural practice, naming, conceptual practice, orientation, and word recognition. The total score ranges from 0 to 70, with lower scores representing milder disease.

SECONDARY OUTCOMES:
Alzheimer's Disease Assessment Scale-Cognitive section(ADAS-cog) | The variations relative to the baseline in the experimental group and the control group after 13 weeks of treatment.
  The comparison of the change values from baseline of ADAS-cog after 13 weeks of treatment between the experimental group and the control group. ADAS-cog assesses seven aspects of cognitive function: word recall, instructions, construction practice, naming, concept practice, orientation, and word recognition. The total score ranges from 0 to 70 points, with lower scores representing a milder condition.
Comparison of the variations in blood ketone values relative to baseline in both groups during the treatment period | During the 26-week treatment course of the experimental group and the control group.
  This measure compares the variations in blood ketone levels relative to the baseline between the experimental group and the control group during the treatment period. It also examines the influence of blood ketone levels on cognitive function; higher blood ketone levels are associated with improved cognitive function and therapeutic efficacy.
Alzheimer's Disease Co-operative Study Activities of Daily Living (ADCS-ADL) | Changes relative to baseline in both groups after 13 weeks and 26 weeks of treatment .
  The comparison of the changes in ADCS-ADL values from the baseline between the experimental group and the control group after 13 and 26 weeks of treatment. The ADCS-ADL is a scale encompassing 23 items, with a total score ranging from 0 to 78. A lower score indicates a higher severity of impairment.
Therapeutic efficacy (evaluated by ADAS-cog) of the Ketogenic Diet (JT821) combined with different drugs after 13 and 26 weeks of treatment | The changes relative to the baseline in both groups after 13 weeks and 26 weeks of treatment.
  The differences in therapeutic efficacy (evaluated by ADAS-cog) of the Ketogenic Diet (JT821) combined with different drugs for the treatment of Alzheimer's disease after 13 and 26 weeks of treatment.
Mini-Mental State Examination (MMSE) | Changes relative to baseline in both groups after 13 weeks and 26 weeks of treatment
  The comparison of the changes in MMSE scores between the experimental and control groups after 13 and 26 weeks of treatment, MMSE tests cognitive function in five areas: orientation, registration, attention and calculation, recall, and language. It consists of 11 questions, with total score ranging from 0-30 points. Lower score indicate greater cognitive impairment.
Quality of Life Alzheimer's Disease（QOL-AD） | Changes relative to baseline in both groups after 13 weeks and 26 weeks of treatment.
  The comparison of the changes in QOL-AD values from baseline between the experimental and control groups after 13 and 26 weeks of treatment. The QOL-AD consists of 13 items, each scored from 1 to 4. For item 7, concerning marital status, if the patient is unmarried, the assessment should be conducted with the closest person available. The overall score ranges from 13 to 54 points, with higher score indicating better the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Jia, Dr., Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Capital Medical University Xuanwu Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No